CLINICAL TRIAL: NCT02589184
Title: Effects on Shoulder Pain of Simulated Hyper-gravity During Rehabilitation Exercises
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics reason at the data collection site
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal investigator, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-IRB-20150818006A
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Shoulder Pain
Keywords: balance, postural; postural equilibrium; pain scale; range of motion
MeSH Terms: conditions — Shoulder Pain | interventions — Hypergravity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- hypergravity WITH isometric load (Experimental): Patient performing rehabilitation exercises under hypergravity as well as loaded isometric squats
  Interventions: Other: Hypergravity; Other: isometric load
- hypergravity WITHOUT isometric load (Experimental): Patient performing rehabilitation exercises under hypergravity
  Interventions: Other: Hypergravity
- normal gravity WITH isometric load (Experimental): Patient performing rehabilitation exercises under normal gravity as well as loaded isometric squats
  Interventions: Other: isometric load; Other: normal gravity
- normal gravity WITHOUT isometric load (Active Comparator): Patient performing rehabilitation exercises under normal gravity
  Interventions: Other: normal gravity

INTERVENTIONS:
Other: Hypergravity — the rubber bands attached to the waist belt are tighten to simulate extra gravity during every exercise the subject performs while standing
  Arms: hypergravity WITH isometric load; hypergravity WITHOUT isometric load
Other: isometric load — at the end of the therapy session the subject will perform 2 sets of one minute each of a 33% squat under load
  Arms: hypergravity WITH isometric load; normal gravity WITH isometric load
Other: normal gravity — the rubber bands attached to the waist belt are NOT tighten so the subject performs the exercises in normal gravity
  Arms: normal gravity WITH isometric load; normal gravity WITHOUT isometric load

SUMMARY:
Determine if adding "extra-gravity" (sustained increase in vertical loading) during standard rehabilitation exercises has a beneficial effect on pain reduction in subjects suffering from shoulder pain of different origin.

DETAILED DESCRIPTION:
Standard rehabilitation protocols will be used with every subject, depending on the cause of their shoulder pain. The treating clinician will determine the appropriate therapy protocol for each subject.

During the treatment sessions, subjects will wear a very comfortable waist belt attached with rubber band to anchor points on the ground (the rubber bands will be tighten to simulate the extra-gravity).

Upon enrollment, the treating clinician will randomly assign the subject to one of four groups depending on the type of loading and exercise typology.

The hyper-gravity will be simulated as an additional 50% of subject's body weight.

The frequency and duration of each therapy session will be determined by the treating clinician (usually 45 minutes of therapy twice a week for 4 weeks).

Before, after and 24h post therapy session, the subject will grade the pain level using a numeric pain scale (0 no pain; 10 unbearable pain requiring pain medication).

As part of the rehabilitation therapy procedure, subjects will undergo shoulder range of motion evaluations (done by a trained clinician in approximately 3 minutes) and Computer Dynamic Posturography (CDP) testing on a 4" tall foam cushion with eyes closed (PSEC test - less than 1 minute of testing) before and after each therapy session.

Subjects will complete the DASH and TOSSA questionnaires (the total amount of time required to complete these assessment is ~20 minutes), and will be tested using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol (the subjects will be required to stand on a hard or compliant surface (a 4" tall foam cushion of known mechanical properties) in a comfortable posture, feet shoulder width, with eyes open or closed, head straight and arms to the side and free to move, gazing forward, and breathing normally, less than 2 minutes testing time) at the time of enrollment and at the end of the 4 week therapy program.

Subjects will be asked to come back for two more evaluations (questionnaires, range of motion assessment, and CDP testing) one month and three months after the end of the 4 week therapy program to identify possible long term effects of the "hyper-gravity/accentuated vertical loading" therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of shoulder pain (potentially including rotator cuff pathology, impingement, bursitis, SLAP tear)

Exclusion Criteria:

* adhesive capsulitis, fracture, dislocation, inflammatory arthritis, cancer, ligament disruption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain level | three months
  The patient will grade the pain level using a numeric pain scale (0 no pain; 10 unbearable pain requiring pain medication).
  Changes will be assessed between baseline (before therapy sessions) and three month post therapy. It will be used to investigate if there is any statistical difference between the different therapies.

SECONDARY OUTCOMES:
Changes in Stability Score | three months
  The Stability Score is calculated as percentage ratio of the actual sway and the theoretical limit of stability.
  Changes will be assessed between baseline (before therapy sessions) and three month post therapy. It will be used to investigate if there is any statistical difference between the different therapies.
Changes in shoulder range of motion | three months
  It is measured as shoulder abduction through "Scaption Range", external / internal rotation in abduction at 90 degrees, and single arm overhead press motion.
  Changes will be assessed between baseline (before therapy sessions) and three month post therapy. It will be used to investigate if there is any statistical difference between the different therapies.
Changes in Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure | three months
  A 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb.
  Changes will be assessed between baseline (before therapy sessions) and three month post therapy. It will be used to investigate if there is any statistical difference between the different therapies.
Test of Sustained Selective Attention (TOSSA) | three months
  An 8-minute computerized auditory sustained attention test. Changes will be assessed between baseline (before therapy sessions) and three month post therapy. It will be used to investigate if there is any statistical difference between the different therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (2):
- United States (2):
  - FIFE Therapy, Savannah, Georgia
  - Optim Orthopedics - DeRenne, Savannah, Georgia